CLINICAL TRIAL: NCT06830031
Title: A Phase 1 Study of C402-CD19-CAR, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Targeting CD19 in Subjects With Relapsed or Refractory Large B-cell Lymphoma
Brief Title: Clinical Study of C402-CD19-CAR Treatment in Subjects With Relapsed or Refractory B-cell Lymphoma
Acronym: C402
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Exuma Biotechnology Ltd. (Industry)
Collaborators: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C402-001
Record Dates: First submitted 2025-02-06; First posted 2025-02-17 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diffuse Large B-cell-lymphoma; DLBCL, Nos Genetic Subtypes; Follicular Lymphoma Grade 3B; PMBL; HGBL With MYC and BCL2 and/or BCL6 Rearrangements; HGBL, Nos
Keywords: autologous fast CAR-T; CD19; B cell lymphoma; subcutaneous injection; without lymphodepletion
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Pyloric Stenosis, Hypertrophic; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C402-CD19-CAR (Experimental): To determine the safety, tolerability, dose-limiting toxicities (DLT) and maximum tolerated dose (MTD) of C402-CD19-CAR cell therapy in patients with relapsed or refractory large B cell lymphoma.
  Dose cohorts:
  * Dose level 1: 0.3x105 CD19 CAR positive cells/kg body weight, subcutaneous injection
  * Dose level 2: 1 x105 CD19 CAR positive cells/kg body weight, subcutaneous injection
  * Dose level 3: 3 x105 CD19 CAR positive cells/kg body weight, subcutaneous injection
  Interventions: Biological: C402-CD19-CAR

INTERVENTIONS:
Biological: C402-CD19-CAR — Enrolled subjects will undergo apheresis to acquire peripheral blood mononuclear cells. C402-CD19-CAR will be generated from the subject's autologous T cells modified from the apheresis product. After C402-CD19-CAR production and product release, subjects will be administered with a single dose of C402-CD19-CAR via subcutaneous injection.

SUMMARY:
This study is to investigate the safety and tolerability of C402-CD19-CAR treatment in subjects with relapsed or refractory large B-cell lymphoma and further determine the recommended Phase 2 dose of C402-CD19-CAR.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase 1 clinical study of C402-CD19-CAR cell therapy, to evaluate the safety, tolerability, efficacy of C402-CD19-CAR in subject with relapsed or refractory large B cell lymphoma.

Subjects that meet inclusion criteria with positive CD19 (IHC ≥50% tumor cells or FACS ≥70% tumor cells) will receive C402-CD19-CAR treatment according to the modified 2+3+3 dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

Must meet all the following inclusion criteria:

1. Male or female 18-75 years (inclusive);
2. Patients can understand this study and capable of providing informed consent;
3. Patients with willingness to be in the study and comply with the study visit procedures and other protocol requirements;
4. Diagnosed with CD19-positive large B-cell lymphoma (LBCL) based on cytology or histology according to the WHO 2016 standards, including diffuse large B-cell lymphoma not otherwise specified (DLBCL-NOS), grade 3b follicular lymphoma (FL), transformed diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma (PMBL), high-grade B-cell lymphoma (HGBL) with MYC, BCL-2, and/or BCL-6 rearrangements, and high-grade B-cell lymphoma not otherwise specified (HGBL-NOS). For CD19 expression status, subjects with a clear past record of tumor histological diagnosis as CD19-positive (within 6 months prior to screening with no CD19-related treatment in the last 6 months) and tumors showing CD19-positive lymphoma levels ≥ 50% by IHC or CD19-positive lymphoma levels ≥ 70% by flow cytometry. If there is no previous CD19 tumor testing or the result is over 6 months prior to screening, a new tumor pathology sample must be provided or re-collected for CD19-positive diagnosis by the institution, with IHC showing CD19-positive lymphoma levels ≥ 50% or flow cytometry showing CD19-positive lymphoma levels ≥ 70%.
5. For refractory or relapsed large B-cell lymphoma subjects, must have received at least anthracycline-based therapy and rituximab (or other CD20-targeted drugs, excluding CD20-negative cases). If previously treated with R-CHOP or other CD20-targeted therapy, the best treatment outcome prior to relapse must have been complete remission (CR). Subjects should meet the criteria for relapse, progression, or failure after second-line therapy; or relapse after autologous hematopoietic stem cell transplantation (auto-HSCT). If the subject has undergone previous auto-HSCT, the best treatment outcome prior to relapse must have been CR, and the relapse should occur more than 12 months after the previous treatment. (Refractory is defined as the best response to the most recent treatment being disease progression or stable disease after at least 2 cycles of the last-line therapy).
6. According to the 2014 Lugano Treatment Response Assessment Criteria, at least one measurable tumor lesion should be present (lesions can be measured with PET results; lymph node lesions [long axis LDi > 15mm] or extra nodal lesions [long axis LDi > 10mm]);
7. Expected survival time greater than 12 weeks;
8. ECOG score of 0-1;
9. Able to establish an intravenous route for PBMC collection, meeting the following hematologic parameters before screening: Hemoglobin ≥ 80 g/L, absolute neutrophil count ≥ 1.0 × 10^9/L, platelet count ≥ 75 × 10^9/L, lymphocyte count ≥ 0.5 × 10^9/L (if using bone marrow stimulants or blood transfusion, a washout period of 7 days is required; for granulocyte colony-stimulating factor [G-CSF] or granulocyte-macrophage colony-stimulating factor [GM-CSF], a washout period of 4 weeks or 5 half-lives is required);
10. Liver and kidney function, as well as heart and lung function, should meet the following requirements:

    1. Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (using the Cockcroft-Gault formula);
    2. Ejection fraction ≥ 50%, with no clinically significant pericardial effusion or pleural effusion detected;
    3. Oxygen saturation ≥ 92% without oxygen support;
    4. Total bilirubin ≤ 1.5 × ULN (for patients with Gilbert's syndrome or lymphoma involving the liver, ≤ 3 × ULN);
    5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN;
    6. Fibrinogen ≥ 1.0 g/L; activated partial thromboplastin time ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN;
11. No more than 1 month prior to screening, the subject must have participated in another interventional clinical study and recovered to a severity level of ≤ 1 for any treatment-related adverse events.

Exclusion Criteria:

1. History of receiving allogeneic hematopoietic stem cell transplantation, adoptive cell therapy (such as CAR-T therapy), or other gene-modified cell therapies;
2. Any active central nervous system (CNS) involvement (including symptomatic and asymptomatic), or a history of CNS disease (such as epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar disorders, or any autoimmune diseases involving the CNS);
3. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA positivity, or subjects with HBV titers above the upper limit of the normal range for the study center; positive for hepatitis C virus (HCV) antibody and peripheral blood HCV RNA positivity; positive for cytomegalovirus (CMV) DNA; positive for human immunodeficiency virus (HIV) antibody; positive for syphilis test;
4. Any unstable systemic disease, including but not limited to unstable angina, cerebrovascular accident or transient ischemic attack (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), active bleeding, severe arrhythmias requiring drug treatment, liver, kidney, or metabolic disorders;
5. Presence of malignant tumors other than large B-cell lymphoma, except for cured non-melanoma skin cancer, carcinoma in situ of the cervix, localized prostate cancer, superficial bladder cancer, ductal carcinoma in situ, and other cancers with a disease-free survival of more than 5 years;
6. Presence of gastric lymphoma, bulky disease, a history of CD19+ leukemia, or active autoimmune diseases (e.g., systemic lupus erythematosus, Sjögren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, Hashimoto's thyroiditis, etc.);
7. Presence of uncontrolled active infections requiring treatment (e.g., sepsis, bacteremia, fungemia, viremia) (mild urinary tract infections or upper respiratory tract infections are exceptions), with the exception of prophylactic anti-infection treatment (for bacterial, fungal, viral infections, etc.);
8. Subjects who have received systemic steroid treatment within 2 weeks before PBMC collection and are determined by the investigator to require long-term systemic steroid treatment during the treatment period (except for inhaled, local application, or physiological replacement doses [hydrocortisone ≤7 mg·d-1 or equivalent prednisone ≤5 mg·d-1 or dexamethasone ≤0.5 mg·d-1]);
9. Subjects who have received anti-tumor treatment within 8 weeks or 5 half-lives (specific medications need to be assessed in detail) before PBMC collection, including chemotherapy, CD20-targeted therapy, etc.; local radiotherapy within 12 weeks;
10. Subjects who have used granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 4 weeks before PBMC collection or within at least 5 half-lives (whichever is shorter);
11. Subjects who have received alendronate treatment within 6 months before PBMC collection, or who have received fludarabine, cladribine, or bendamustine treatment within 3 months before PBMC collection;
12. Subjects who have undergone major surgery within 4 weeks prior to screening (as defined by "Clinical Application Measures of Medical Technology" and "Grade 3 and 4 surgeries") or who have not fully recovered from any previous invasive procedure;
13. Subjects who have received a live vaccine within 28 days before PBMC collection;
14. Pregnant or breastfeeding women, or those who plan to become pregnant during the treatment period or within 2 years after treatment, or male subjects whose partners plan to become pregnant within 2 years after male subject's cell injection;
15. Subjects whom the investigator deems unsuitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2026-03-09 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
MTD (maximum tolerated dose) of C402-CD19-CAR | 28 days following injection
  To evaluate the DLT (dose limiting toxicities), attributed to C402-CD19-CAR per cohort and determine the RP2D (recommended phase 2 dose).
AE (Adverse Event), AESI (Adverse Event of Special Interest), SAE (Severe Adverse Event) | up to 2 years post injection
  The incidence, severity and duration of AE, AESI and SAE as determined by NCI-CTCAE v5.0

SECONDARY OUTCOMES:
ORR (Objective Response Rate) | up to 2 years post injection
  ORR and best overall response (BOR) of subjects with PR (partial response) and CR (complete response) as determined by local investigator using Lugano 2014
DOR (Duration of response) | up to 2 years post injection
  The duration of time from record of response to first progression of disease or death as determined by Lugano 2014
PFS (Progression free survival) | up to 2 years post injection
  The duration of time from treatment to first progression of disease as determined by Lugano 2014
DCR (Disease control rate) | up to 2 years post injection
  The proportion of subjects with CR (complete response), PR (partial response) or SD (stable disease lasting over 6 months) to total number of patients treated as determined by local investigator using Lugano 2014
OS (Overall Survival) | up to 15 years post injection
  The time from the start of treatment to the occurrence of death due to any cause
PK (Pharmacokinetics): AUCinf | up to 2 years post injection
  Calculate AUCinf: area under the blood concentration-time curve extrapolated to infinity
PK: AUC(0-t) | up to 2 years post injection
  calculate AUC(0-t): the AUC from time 0 to the last measurable concentration that represents the observed exposure to a drug
PK: AUC0-28d | up to 2 years post injection
  calculate AUC0-28d: the area under the concentration-time curve from day 0 to day 28
PK: AUC0-90d | up to 2 years post injection
  Calculate AUC0-90d: the area under the concentration-time curve from day 0 to day 90
PK: Cmax | up to 2 years post injection
  Calculate Cmax: the highest concentration of the drug in the blood
PK: half-life | up to 2 years post injection
  Calculate half-life: the time it takes for the amount of the drug's active substance in your body to reduce by half
PK: Tmax | up to 2 years post injection
  Calculate Tmax: the time it takes for the drug to reach the maximum concentration after administration of a drug that needs to be absorbed
PK: MRT | up to 2 years post injection
  Calculate MRT (Mean Residence Time): the average time a molecule spends in a system before being removed)
Concentration of cytokines | up to 2 years post injection
  Test serum concentration of IL-2、IL-4、IL-6、IL-10、IFN-γ、TNF-α before and post C402-CD19-CAR treatment
Concentration of Anti-Drug Antibody | up to 2 years post injection
  Test antibodies that form in response to the administration of C402-CD19-CAR

OTHER OUTCOMES:
Correlation between PK, cytokine concentration and efficacy | up to 2 years post injection
  Calculate the correlation between PK data, cytokine concentration with efficacy parameters (PFS, OS, ORR, DCR, DOR)
B cell count | up to 2 years post injection
  Test B cell count and the subsets percentage in blood before and post C402-CD19-CAR treatment
RCL (replication-competent lentivirus) test | up to 15 years post injection
  Test VSVG copies/μg gDNA in blood after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Liang Huang, MD, Principal Investigator — Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu W, Liu J, Song Y, Zeng X, Wang X, Mi L, Cai C, Wang L, Ma J, Zhu J; Union for China Leukemia Investigators of the Chinese Society of Clinical Oncology; Union for China Lymphoma Investigators of the Chinese Society of Clinical Oncology. Burden of lymphoma in China, 2006-2016: an analysis of the Global Burden of Disease Study 2016. J Hematol Oncol. 2019 Nov 19;12(1):115. doi: 10.1186/s13045-019-0785-7. PMID 31744509
- [Result] Liu W, Liu J, Song Y, Wang X, Mi L, Cai C, Zhao D, Wang L, Ma J, Zhu J. Burden of lymphoma in China, 1990-2019: an analysis of the global burden of diseases, injuries, and risk factors study 2019. Aging (Albany NY). 2022 Apr 10;14(7):3175-3190. doi: 10.18632/aging.204006. Epub 2022 Apr 10. PMID 35398840
- [Result] Zahid U, Akbar F, Amaraneni A, Husnain M, Chan O, Riaz IB, McBride A, Iftikhar A, Anwer F. A Review of Autologous Stem Cell Transplantation in Lymphoma. Curr Hematol Malig Rep. 2017 Jun;12(3):217-226. doi: 10.1007/s11899-017-0382-1. PMID 28478586
- [Result] Li X, Ding Y, Zi M, Sun L, Zhang W, Chen S, Xu Y. CD19, from bench to bedside. Immunol Lett. 2017 Mar;183:86-95. doi: 10.1016/j.imlet.2017.01.010. Epub 2017 Jan 30. PMID 28153605